CLINICAL TRIAL: NCT02817490
Title: Evaluation of an Education Program for Patients With Hypermobility Type Ehlers-Danlos Syndrome
Brief Title: Patient Education Program and Ehlers-Danlos Syndrome
Acronym: PREDUSED
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D21775
Record Dates: First submitted 2016-06-24; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Hypermobility Type Ehlers-Danlos Syndrome
Keywords: hypermobility; Ehlers-Danlos Syndrome; patient education program
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3; Ehlers-Danlos Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with hypermobility type Ehlers-Danlos Syndrome: Patients with hypermobility type Ehlers-Danlos Syndrome participating to one out of the three patient education sessions included in the study.
  Interventions: Other: patient education program
- Caregivers: Caregivers participating to one out of the three patient education sessions included in the study.
  Interventions: Other: patient education program

INTERVENTIONS:
Other: patient education program — The PREDUSED patient education program aims to make the patient actor of his pathology by providing him a "box of therapeutic tools" in order to: improve his knowledge of the disease, improve the management of pain, fatigue and episodes of instability; learn to communicate about the disease; set realistic goals.
  The program includes theoretical information, practical cases, and discussions between participants and professionals.
  It is the first patient education program in France for the patients with hypermobility type Ehlers-Danlos Syndrome. It is proposed two times a year. Six patients can participate at each session.

SUMMARY:
The Ehlers-Danlos Syndrome (SED) comprises a group of clinically and genetically heterogeneous, inherited connective tissue diseases. The hypermobility type is the most frequent. It is characterized by a generalized joint hypermobility and a hyperextension skin.

Chronic pain syndrome is often present. Its psychological impact can be significant (anxiety, depression, impact on the quality of life of the patients). The disease also requires changes and a permanent adaptability (coping). It can lead to feelings of isolation and misunderstanding.

The French association of the Ehlers-Danlos Syndromes and the rehabilitation center of the 'Croix-Rouge Française des Massues' propose a patient education program for the patients with a hypermobility type SED (the PrEduSED program). This education program is open to patients and their caregivers located in France.

The research hypothesis is that the PrEduSED program improves their coping and reduces patient anxiety at 6 months (these are the two clinical criteria on which the PrEduSED could have the most impact, given the results of the first sessions).

ELIGIBILITY:
Inclusion Criteria:

Patients

* adults (>18 years)
* hypermobility type Ehlers-Danlos Syndrome
* participating to one education session during the study period

Caregivers

* adults (>18 years)
* caregivers of patients with hypermobility type Ehlers-Danlos Syndrome
* participating to one education session during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hypermobility type Ehlers-Danlos Syndrome and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Changes in scores obtained on the Coping Strategies Questionnaire-French version (CSQ-F) | Just before the education program (day 0) and 6 months after the education program (month 6)
  The Coping Strategies Questionnaire-French version - CSQ-F measured the pain coping strategies through 21 items.
  It evaluates the behavioral level of the Kirkpatrick model, the degree to which participants apply what they learned during training (level 3)

SECONDARY OUTCOMES:
Changes in Hospital Anxiety And Depression Scale (HAD) | administered just before (day 0) and 6 months after the education program (month 6)
  It contains 14 items. It evaluates the result level of the Kirkpatrick model, the degree to which targeted outcomes occur as a result of the training (level 4)
Changes in a satisfaction questionnaire | administered just after the education program (day 4)
  It evaluates the reaction level of the Kirkpatrick model, the degree to which participants find the training favorable, engaging and relevant (level 1)
Changes in a quiz | administered just before (day 0), after the education program (day 4) and 6 months after
  It evaluates the learning level of the Kirkpatrick model, the degree to which participants acquire the intended knowledge, skills, attitude (level 2)
Changes in a Goal Attainment Scaling (GAS) | administered just before (day 0), after the education program (day 4)
  It evaluates the learning level of the Kirkpatrick model, the degree to which participants acquire the intended knowledge, skills, attitude (level 2)

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine TOUZET, MD, Principal Investigator — Pôle Information Médicale Evaluation Recherche - Hospices Civils de Lyon
Locations (1):
- Pôle Information Médicale Evaluation Recherche - Hospices Civils de Lyon, Lyon, France